CLINICAL TRIAL: NCT01406054
Title: Role of Neuromuscular Training in Reducing Sports Injuries and Improving Fitness Among Chicago Public Elementary and Middle School Students
Brief Title: Neuromuscular Training to Reduce Sports Injuries Among Children and Adolescents
Acronym: KIPP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Principal Investigator, Cynthia LaBella, Attending Physician, Orthopaedic Surgery and Sports Medicine, Ann & Robert H Lurie Children's Hospital of Chicago
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB 2011-14570
Record Dates: First submitted 2011-07-28; First posted 2011-07-29 (Estimated); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Leg Injuries
Keywords: athletes; injury prevention; neuromuscular training; public school; physical education; knee; sports; ACL; KIPP
MeSH Terms: conditions — Leg Injuries

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- neuromuscular training (Experimental): subjects in this arm will undergo neuromuscular warm-up exercises before practices and games
  Interventions: Other: neuromuscular exercises
- control (No Intervention): subjects in the control arm will proceed to practice and games without additional neuromuscular warm-up exercises.

INTERVENTIONS:
Other: neuromuscular exercises — neuromuscular exercises delivered as a pre-practice and pre-game warm-up including dynamic stretching, strengthening, and plyometrics.
  Other Names: KIPP
  Arms: neuromuscular training

SUMMARY:
Sports-related injuries are a serious concern for physically active children and adolescents. Previous research, including ours at Chicago public high schools, shows our neuromuscular training program, the Knee Injury Prevention Program (KIPP) reduces sports-related injuries in female athletes by up to 88%. However, KIPP is not well-studied in males or younger age groups. This project aims to determine KIPP's effect on sports-related injuries and physical fitness among 5th-8th grade students in Chicago public schools. The study will take place during the 2011-2013 school years. To measure KIPP's effect on sports injuries, we will recruit 5th-8th grade sports coaches and their athletes, randomize coaches by school into two groups, then train the intervention group to implement a 10-minute KIPP warm-up before practices and games. Control group will perform their usual warm-up. Research assistants will collect athlete participation and injury data from coaches weekly. To determine feasibility of KIPP in PE classes and measure its effect on fitness, we will recruit PE teachers to implement the warm-up in PE classes for a minimum of 10 weeks, and record students' presidential fitness test scores before and after the 10+ weeks. Results of this study will guide strategies for preventing sports-related injuries and improving physical fitness in 5th -8th graders.

DETAILED DESCRIPTION:
PURPOSE OF THE RESEARCH

The long-term goal is to reduce sports-related injuries and improve physical fitness in children and adolescents by incorporating the neuromuscular training program called the Knee Injury Prevention Program (KIPP) into their physical education classes or sports practice routines. This project aims to measure the effectiveness of KIPP in reducing injuries and improving physical fitness among 5th -8th grade boys and girls in Chicago public schools. Specifically, the investigators aim to:

* Train PE teachers and sports coaches for 5th -8th grade students how to incorporate the 10-minute KIPP warm-up into their regular team practices and PE classes.
* Measure the effect of KIPP on sports injury rates.
* Measure the effect of KIPP on PE students' physical fitness.

LITERATURE REVIEW / JUSTIFICATION OF RESEARCH Sports-related injuries are a serious concern for physically active children and adolescents. Treatment costs can be substantial, and the time lost from school and sports can have considerable impact on mental health and academic performance. A handful of studies, including our previous research in CPS high schools, have shown that coach-led neuromuscular training (NMT) programs can reduce the risk for sports-related injuries among female high school athletes by up to 88%. However, few studies of NMT have included athletes under 14 years of age, and none have investigated the protective effect of NMT in sports other than soccer, basketball, volleyball and team handball. NMT includes exercises to strengthen the core and lower extremity muscles, improve balance and agility, and promote safe techniques with landing and pivoting which are the most common sports maneuvers that lead to injury.

In 2006, the investigators researched a coach-led neuromuscular training program called the Knee Injury Prevention Program (KIPP) for female soccer and basketball athletes in CPS high schools and found a statistically significant reduction in lower extremity injuries in the teams using the KIPP warm-up. KIPP should also have beneficial effects on physical fitness; however this has not yet been directly studied.

HYPOTHESES

* Coaches and PE teachers will demonstrate compliance and competency with implementing KIPP exercises into their regular practices/games and PE classes, respectively.
* KIPP training will reduce injuries in school-sponsored sports.
* KIPP training will improve PE students' physical fitness.

PRELIMINARY STUDIES From 2006 to 2007, we researched coach-led KIPP among female soccer and basketball athletes in Chicago Public High Schools and found significant reduction in lower extremity injuries. In 2005, we conducted a trial of pre-season KIPP for female adolescent athletes and found a reduction in subjects' sports-related knee pain pre- vs. post-training.

DESCRIPTION OF RESEARCH APPROACH This will be a cluster-randomized, controlled trial. The Acting Officer for the Office of Student Support and Engagement, the Director of Athletics for Chicago Public Schools (CPS), and the CPS Office of Student Health and Wellness understand and support the project's goals and research methods. CPS has agreed to provide PE teachers and coaches with staff development credits as an incentive to complete the study. The study will be implemented by "study personnel" who are all Lurie Children's-affiliated health care professionals or employees.

ELIGIBILITY:
Inclusion Criteria:

* sports coaches and physical education (PE) teachers for 5th-8th grade students at a CPS school
* 5th-8th grade students/athletes at a chicago public school

Exclusion criteria:

* Not a coach or PE teacher at CPS
* not a 5th-8th grade student at CPS

Ages: 10 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 400 (Actual)
Dates: Start 2011-07 (Actual); Primary Completion 2020-06 (Actual); Study Completion 2021-07 (Actual)

PRIMARY OUTCOMES:
sports-related lower extremity injuries | 0-3 years
  Frequency of injuries

SECONDARY OUTCOMES:
physical fitness as measured by presidential fitness test | 0-3 years

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia LaBella, MD, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago
Locations (1):
- Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois, United States